CLINICAL TRIAL: NCT00393302
Title: HIV Testing in Pregnant Women: An Evaluation of an Opt-Out Strategy in an Ambulatory Care Clinic Setting
Brief Title: HIV Testing in Pregnant Women: Evaluating an Opt-Out Testing Strategy
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Dr. Mark Yudin, Obstetrician/Gynecologist, Research Scientist, St. Michael's Hospital
Other Study IDs: 03-326
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: HIV; AIDS Virus; Pregnancy
Keywords: HIV testing in pregnant women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — HIV Testing; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 & 2: 1. Retrospective chart review: HIV testing rates
  2. Prospective cohort group: HIV testing rates
  Interventions: Procedure: HIV screening in pregnancy

INTERVENTIONS:
Procedure: HIV screening in pregnancy

SUMMARY:
Mother-to-child transmission of HIV is an important but preventable mode of infection. Prevention depends on identifying pregnant women infected with HIV and offering medications during pregnancy which can dramatically decrease the chances of transmission. Currently universal screening of all pregnant women for HIV is recommended in the province of Ontario. Unfortunately the rates of screening are still low: estimates place the average rate at 50% -60%. We believe that rates in our clinic at the Women's Health Care Centre are significantly higher in part because all our patients have a first obstetrical visit. This is an unhurried visit with a trained obstetrical nurse who offers pre-test counselling and explores reasons why patients refuse testing. We hypothesize that with this system, acceptance rates for HIV screening are significantly higher than the provincial average.

DETAILED DESCRIPTION:
We hypothesize that by having a dedicated and unhurried intake visit with a trained obstetrical nurse, pregnant women will be more likely to accept antenatal HIV testing. We further hypothesize that in our obstetrical clinic at the Women's Health Care Centre, the application of a universal opt-out screening policy will result in a testing rate that is higher than the provincial average.

This is a two part study. The first part will be a retrospective chart review while the second part will be a prospective cohort study. All antenatal patients with first visits at our clinic will be included. For the retrospective portion, 537 charts will be reviewed. For the prospective portion, 537 patients will be enrolled prospectively using a data sheet which will be included in all charts starting when the study begins. For both portions, the following information will be obtained:

* presence of HIV test
* result of test
* if test not performed, the reason documented, in any
* if testing refused, the reason for refusal

Additional information that will be obtained includes:

* number of HIV positive pregnant women cared for in our clinic during the study period
* percentage of positive cases
* difference in testing (acceptance) rates between the retrospective and prospective (when data sheet in use) portions of the study.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women attending antenatal intake appointments at the Women's Health Care Centre at St. Michael's Hospital in Toronto, Canada between September 2003 and February 2005.

Exclusion Criteria:

* Any pregnant women obtaining antenatal care at other health care facilities.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All pregnant women attending antenatal intake appointments at the Women's Health Care Centre at St. Michael's Hospital in Toronto, Canada between September 2003 and February 2006.
Sampling Method: Non-Probability Sample
Enrollment: 1074 (Actual)
Dates: Start 2003-09; Primary Completion 2006-01 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Yudin, MD MSc, Principal Investigator — St. Michael's Hospital & the University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Yudin MH, Moravac C, Shah RR. Influence of an "opt-out" test strategy and patient factors on human immunodeficiency virus screening in pregnancy. Obstet Gynecol. 2007 Jul;110(1):81-6. doi: 10.1097/01.AOG.0000267497.39041.06. PMID 17601900